CLINICAL TRIAL: NCT05146284
Title: A Randomized Open-label Phase 2a Study to Assess PXL770 After 12 Weeks of Treatment in Male Subjects With Adrenomyeloneuropathy (AMN) Form of X-linked Adrenoleukodystrophy (X-ALD or ALD)
Brief Title: Study to Assess PXL770 in Subjects With Adrenomyeloneuropathy (AMN) Form of X-linked Adrenoleukodystrophy (X-ALD or ALD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding to initiate the study
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PXL770-011
Record Dates: First submitted 2021-11-16; First posted 2021-12-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Adrenomyeloneuropathy
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — 2-chloro-3-(1-hydroxy-5,6,7,8-tetrahydronaphthalen-2-yl)-6-oxo-5-phenyl-7H-thieno)(2,3-b)pyridin-4-olate potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PXL770 500 mg QD (Experimental)
  Interventions: Drug: PXL770
- PXL770 250 mg BID (Experimental)
  Interventions: Drug: PXL770

INTERVENTIONS:
Drug: PXL770 — Tablet

SUMMARY:
A randomized open-label Phase 2a study to assess the pharmacokinetics and pharmacodynamic parameters of PXL770 after 12 weeks of treatment in male subjects with adrenomyeloneuropathy (AMN).

DETAILED DESCRIPTION:
A randomized open-label Phase 2a study to assess the pharmacokinetics and pharmacodynamic parameters of PXL770 after 12 weeks of treatment in male subjects with adrenomyeloneuropathy (AMN).

There are 3 study periods.

* Screening Visit: within a maximum of 4 weeks prior to the open-label Treatment Period
* Open-label Treatment Period: 12 weeks
* Follow-up Period: 2 weeks after the last intake of the treatment

During the treatment period, VLCFA will be assessed every 4 weeks, to evaluate the kinetics of the effect. NfL will be assessed after 8 and 12 weeks of treatment, and other exploratory biomarkers after 12 weeks of treatment. A follow up period will allow monitoring the subjects' safety as well as the duration of the effect on the 2 main biomarkers (VLCFA and NfL) at 2 and 4 weeks after the drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with either a confirmed diagnosis of AMN by genetic testing (mutation in the ATP binding cassette subfamily D (ABCD1 gene)) or a family history of X-linked adrenoleukodystrophy (ALD) together with an elevation in VLCFA obtained from overnight fasting plasma sample at Screening Visit (V1).
* Age: ≥ 18 to ≤ 65 years at informed consent signature.
* Normal brain magnetic resonance imaging (MRI) or brain MRI showing non-specific abnormalities that can be observed in AMN subjects without signs of cerebral form of ALD (C-ALD). MRI must be performed within 6 months prior to V2. If there is no available brain MRI within this period, a brain MRI must be performed before V2.

Exclusion Criteria:

* Any progressive neurological disease other than AMN.
* Arrested or progressing C-ALD as defined by cerebral lesions (except for non-specific abnormalities that can be observed in AMN subjects).
* Prior receipt of an allogeneic hematopoietic stem cell transplant or gene therapy.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters | 4 week
  Peak plasma concentration (Cmax) for 500mg QD
Pk parameters | 4 week
  Area under the plasma concentration versus time curve (AUC)0-24 for 500mg QD
PK parameters | 4 week
  Cmax for 250mg BID
PK parameters | 4 week
  AUC0-8 for 250mg BID

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers